CLINICAL TRIAL: NCT06953063
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study To Evaluate The Efficacy And Safety Of DA-302168S Tablets In Overweight/Obese Subjects
Brief Title: A Study to Evaluate the Efficacy and Safety of DA-302168S Tablets in Overweight/Obese Subjects
Acronym: DA168
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chendu DIAO Pharmaceutical Group CO., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-CP-DA168-06
Record Dates: First submitted 2025-04-11; First posted 2025-05-01 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Overweight and Obesity
Keywords: Overweight and Obesity; GLP-1
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DA-302168S (Experimental): 5mg dose group：Participants will receive DA-302168S tablets once daily orally, 16weeks.
  10mg dose group：Participants will receive DA-302168S tablets once daily orally, 16weeks.
  20mg dose group：Participants will receive DA-302168S tablets once daily orally, 16weeks.
  30mg dose group：Participants will receive DA-302168S tablets once daily orally, 16weeks.
  Interventions: Drug: DA-302168S
- Placebo of DA-302168S (Placebo Comparator): 5mg dose group：Participants will receive matching placebo tablets orally once daily for 16 weeks.
  10mg dose group：Participants will receive matching placebo tablets orally once daily for 16 weeks.
  20mg dose group：Participants will receive matching placebo tablets orally once daily for 16 weeks.
  30mg dose group：Participants will receive matching placebo tablets orally once daily for 16 weeks.
  Interventions: Drug: Placebo of DA-302168S

INTERVENTIONS:
Drug: DA-302168S — A small molecule GLP-1R agonist tablet, orally administration, once daily，16weeks.
  Arms: DA-302168S
Drug: Placebo of DA-302168S — Matching placebo tablet will be provided
  Arms: Placebo of DA-302168S

SUMMARY:
It is a multicenter, randomized, double-blind, placebo-controlled phase II clinical trial to evaluate the safety and efficacy of DA-302168S tablets in overweight and obese adults.

DETAILED DESCRIPTION:
The goal of the study is to assess how DA-302168S tablets affect the bodyweight when used once daily in obese or overweight adult participants. Qualified participants will be randomly assigned to one of five groups using a computerized system. Following the screening period to confirm eligibility up to 2-weeks, the study will consist of a treatment period will be 16 weeks, followed by an approximate 2-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age range:18-75 years old (inclusive),regardless of gender;
2. BMI requirements at screening:obese patients, BMI >28 kg/m2 with or without comorbidities; or, overweight patients, BMI =24.0 kg/m2 but 28 kg/m2 with at least one；
3. Weight change (weight change [maximum weight-minimum weight] /maximum weight;based on subject self-report)did not exceed 5%during the 3 months before screening under diet and exercise control;

Exclusion Criteria:

1. Secondary obesity: including obesity previously diagnosed as endocrine disease or caused by single gene mutation (including but not limited to hypothalamic obesity, pituitary obesity, Cushing's syndrome, hypothyroidism, islet cell tumor, acromegaly, hypogonadism, polycystic ovary syndrome, etc.) or drug-induced obesity (such as glucocorticoids, tricyclic antidepressants, atypical antipsychotics, etc.)
2. Those who have undergone weight loss surgery in the past (except for acupuncture weight loss, liposuction and abdominal fat removal surgery one year before screening), or plan to undergo surgery for obesity during the study period, such as gastric bypass, gastric banding, etc.;
3. The patient has clinically cardiovascular and cerebrovascular diseases, including but not limited to the following cardiovascular and cerebrovascular diseases or conditions within 6 months before signing the ICF: a. Unstable angina pectoris; b. Heart failure (New York Heart Association heart function grade III or IV); c. Myocardial infarction; d. Coronary artery bypass grafting or percutaneous coronary intervention; e. Uncontrolled severe arrhythmia, such as sick sinus syndrome, second or third degree atrioventricular block, etc.; f. Cerebrovascular accident, such as cerebral infarction, transient ischemic attack, etc.
4. Those who had acute pancreatitis 3 months before signing the ICF, or had a history of chronic pancreatitis or pancreatic injury, which may be high-risk factors for pancreatitis;
5. Individuals who have experienced acute cholecystitis in the 3 months prior to signing the ICF, or have cholecystitis/cholangitis/bile duct stones/multiple gallstones at screening, or have been assessed by researchers as having gallbladder-related diseases that may lead to a high incidence of cholecystitis during screening;
6. Sufering from any malignant tumor within 5 years before signing the ICF (except cured basal cell carcinoma of the skin or carcinoma in situ of the cervix);
7. A history or family history of medullary thyroid cancer, thyroid C-cell hyperplasia, or multiple endocrine neoplasia type 2;
8. Patients with a history of thyroid dysfunction who still require medication during screening, or with clinically significant abnormal thyroid function results during screening, or with thyroid nodules assessed by researchers as having safety risks during screening.;
9. Those who have experienced severe hypoglycemia or repeated symptomatic hypoglycemia (≥2 times within half a year) in the past (severe hypoglycemia is defined as: severe events accompanied by changes in consciousness and/or body, hypoglycemia that requires help from others);
10. Those with a specific allergy history that, as assessed by the investigator, will significantly affect the safety of the subjects (such as asthma, urticaria, eczema, etc.) or allergic constitution, or those who are allergic to any component of the trial drug or preparation, or those who are allergic to other glucagon-like peptide-1 receptor agonist (GLP-1RA) drugs or drugs with a glucagon-like peptide-1 (GLP-1) receptor stimulating mechanism;
11. HbA1c ≥ 6.5%, or FPG ≥ 7.0 mmol/L or ≤ 3.9 mmol/L at screening, or patients previously diagnosed with type 1 diabetes, type 2 diabetes, or other special types of diabetes (according to the diabetes diagnosis and classification criteria issued by the World Health Organization [WHO] in 2019;
12. Those with a history of moderate to severe depression, anxiety, or severe mental illness, or those with a depression screening scale (PHQ-9) score ≥ 15 at screening (see Appendix 3 for details); 13 Have a history of dysphagia or any gastrointestinal disease that affects drug absorption, including but not limited to gastrectomy or any intestinal resection, severe gastrointestinal disease, clinically obvious gastric emptying abnormalities, etc.;

14.People who are lactose intolerant (for example, those who have had diarrhea after drinking milk within the shelf life); 15.During screening, the clinical laboratory test (local laboratory) results showed any of the following abnormalities (rechecked and confirmed once within 1 week if necessary): 1) hemoglobin <100 g/L for females and <110 g/L for males; alanine aminotransferase (ALT) ≥2.0×upper limit of normal (ULN); 2) aspartate aminotransferase (AST) ≥2.0×ULN; 3) total bilirubin (TBIL) ≥1.5×ULN; 4) blood amylase or blood lipase >1.5×ULN; 5) calcitonin ≥1.0×ULN; 6) estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 [Chronic Kidney Disease Epidemiology Institute (CKD-EPI) formula, see Appendix 4 for details]; 7) TG >500 mg/dl (5.65 mmol/L); 8) thyroid stimulating hormone >6 mIU/L or <0.4 mIU/L; 16.Uncontrolled hypertension at screening: systolic blood pressure ≥160 mmHg, or diastolic blood pressure ≥100 mmHg; 17.During screening, 12-lead ECG examinations were performed three times in the supine position at rest, and the average corrected QT interval (corrected according to Fridericia's formula, see Appendix 5 for details) obtained from the three measurements was >450 msec; 18.Those with a history of drug abuse in the past five years or who had used drugs in the three months before screening; 19 Received any GLP-1 RA before screening (including GLP-1R agonists, GLP-1R related multitarget agonists, or compound preparations containing GLP-1R agonists, etc.); 20.Female subjects who are pregnant or breastfeeding, or have a positive pregnancy test; 21.Drugs that may affect body weight were used within 3 months before screening, including: dipeptidyl peptidase-4 (DPP-4) inhibitors, sodium-glucose co-transporter-2 (SGLT-2) inhibitors, insulin, metformin, insulin secretagogues, or thiazolidinedione (TZD) and other hypoglycemic drugs; any approved or unapproved weight loss drugs, such as orlistat, Lorcaserin, phentermine/topiramate, naltrexone/bupropion, etc.) or Chinese herbal medicines, health products, meal replacements, etc. that affect body weight; systemic steroid hormones (intravenous, oral or intra-articular); tricyclic antidepressants, antipsychotics or anti-epileptic drugs (such as imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid, valproic acid derivatives, lithium salts), etc.; Note: Except for those who have used systemic hormones for less than 7 days cumulatively or continuously; 22.Active autoimmune diseases (such as lupus, rheumatoid arthritis), who may be treated with systemic glucocorticoids during the study period as determined by the investigator; 23.Participants who have participated in clinical trials of other drugs within the previous 3 months and received the investigational drug (excluding those who received a placebo); 24. Those who donated blood or lost ≥400 mL of blood, received blood transfusion, or used blood products within 3 months before screening; 25 Heavy smokers or those who smoked ≥5 cigarettes per day on average within 3 months before screening; 26 Heavy drinkers or regular drinkers within 3 months before screening, that is, drinking more than 14 standard units of alcohol per week (1 unit of alcohol = 360 mL of beer or 45 mL of 40% alcohol liquor or 150 mL of wine); 27 Patients with positive results in any of the tests for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab)or Treponema pallidum antibody (TP-Ab); patients with hepatitis B who are HBsAg negative but are undergoing antiviral treatment; 28 The investigator believes that there are other factors that may affect the evaluation of relevant indicators of the effectiveness and safety of this study and make the subject unsuitable for participation in this clinical trial (including but not limited to the investigator's judgment that the subject's compliance is poor, or the subject lives too far away and cannot be followed up as scheduled, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
percentage change in body weight | From baseline (week1) to week16
  percentage-point

SECONDARY OUTCOMES:
Proportion of subjects with weight decrease ≥ 5% | From baseline (week 1) to week 16
  percentage-point
Adverse events, including treatment-emergent adverse events (TEAEs), serious adverse events (SAEs) | From baseline (week 1) to week 18
  Count of events
Proportion of subjects with weight decrease ≥ 10% | From baseline (week 1) to week 16
  percentage-point
Absolute change in body mass index (BMI) | From baseline (week 1) to week 16
  measured in kg/m^2
Absolute change in waist circumference | From baseline (week 1) to week 16
  measured in cm
Absolute change in hip circumference | From baseline (week 1) to week 16
  measured in cm
Change in blood lipid profiles (TC, TG, LDL-C, and HDL-C) | From baseline (week 1) to week 16
  measured in mmol/L
Change in fasting plasma glucose (FPG) | From baseline (week 1) to week 16
  measured in mmol/L
Change in HbA1c (glycated haemoglobin) | From baseline (week 1) to week 16
  percentage-point
Change in fasting insulin | From baseline (week 1) to week 16
  measured in μIU/mL
Change in HOMA-IR | From baseline (week 1) to week 16
  point
Blood pressure (systolic and diastolic) | From baseline (week 1) to week 16
  measured in mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No